CLINICAL TRIAL: NCT00679367
Title: A Phase II Trial of MRD (Melphalan, Lenalidomide and Dexamethasone) for Patients With AL Amyloidosis
Brief Title: Melphalan, Lenalidomide, and Dexamethasone in Treating Patients With Primary Systemic Amyloidosis
Acronym: MRD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Vaishali Sanchorawala, Principal Investigator, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000595759; RV-AMYL-PI-0219 (Other Grant/Funding Number: Celgene); BUMC-H-26320 (Other: Boston University Medical Center IRB)
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2016-12

CONDITIONS: Multiple Myeloma
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Dexamethasone; Calcium Dobesilate; Lenalidomide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melphalan Revlimid and Dexamethasone (Experimental): Melphalan Lenalidomide Dexamethasone
  Interventions: Drug: dexamethasone; Drug: lenalidomide; Drug: melphalan

INTERVENTIONS:
Drug: dexamethasone — 40 mg once weekly
  Other Names: Decadron
Drug: lenalidomide — 10 mg/day D1-21
  Other Names: revlimid, cc-5013
Drug: melphalan — 5 mg/m2 D1-4
  Other Names: alkeran

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan and dexamethasone, work in different ways to stop the growth of abnormal plasma cells, either by killing the cells or by stopping them from dividing. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop the abnormal plasma cells from growing. Giving melphalan together with lenalidomide and dexamethasone may be an effective treatment for primary systemic amyloidosis.

PURPOSE: This phase II trial is studying the side effects and how well giving melphalan together with lenalidomide and dexamethasone works in treating patients with primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the tolerability and safety of melphalan, lenalidomide, and dexamethasone, in terms of toxicity, in patients with primary systemic amyloidosis.
* To determine the hematologic response rate in patients treated with this regimen.

Secondary

* To assess organ response in patients treated with this regimen.

OUTLINE: Patients receive oral lenalidomide once daily on days 1-21, oral melphalan once daily on days 1-4, and oral dexamethasone once on days 1, 8, 15, and 22. Treatment repeats every 28 days for up to 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 3 months until disease progression and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Diagnosis of primary systemic amyloidosis

PATIENT CHARACTERISTICS:

* Not pregnant
* Negative pregnancy test
* Able to tolerate an anticoagulation regimen (e.g., 325 mg of aspirin per day, therapeutic warfarin, or low molecular weight heparin)

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy

  * Permanent or stable side effects/changes allowed
* Prior chemotherapy, thalidomide, lenalidomide, or steroids for amyloidosis allowed
* More than 4 weeks since prior and no other concurrent cytotoxic chemotherapy or radiotherapy

Exclusion Criteria:

* No secondary or familial amyloidosis
* No multiple myeloma (≥ 30% plasma cells in bone marrow biopsy or lytic bone lesions)
* No prior cumulative doses of oral melphalan > 200 mg
* No more than one prior course of high-dose melphalan with stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchorawala V, Patel JM, Sloan JM, Shelton AC, Zeldis JB, Seldin DC. Melphalan, lenalidomide and dexamethasone for the treatment of immunoglobulin light chain amyloidosis: results of a phase II trial. Haematologica. 2013 May;98(5):789-92. doi: 10.3324/haematol.2012.075192. Epub 2012 Nov 9. PMID 23144200

RESULTS

PARTICIPANT FLOW:
Groups:
- Melphalan Revlimid and Dexamethasone: Melphalan Lenalidomide Dexamethasone
  dexamethasone: 40 mg once weekly
  lenalidomide: 10 mg/day Days 1-21
  melphalan: 5 mg/m2 Days 1-4
Period: Overall Study
Arm/Group | Melphalan Revlimid and Dexamethasone
Started | 16
Completed | 4
Not Completed | 12
Not completed — Adverse Event | 7
Not completed — inability to swallow oral drugs | 1
Not completed — Lack of Efficacy | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Melphalan Revlimid and Dexamethasone
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Gender [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hematologic Response
Description: Complete hematologic response: Absence of detectable monoclonal protein in serum or urine by immunofixation electrophoresis, bone marrow biopsy with less than 5% plasma cells without clonal dominance of kappa or lambda isotype, and normal serum free light chain assay.
  Partial hematologic response: Amyloid patients have highly individualized measures of disease burden. For patients with detectable and quantifiable monoclonal marrow plasmacytosis, a reduction of 50% or more in plasma cells as a percentage of nucleated bone marrow cells. For patients with a detectable monoclonal peak on serum or urine protein electrophoresis, a reduction in the peak height of 50% or more. For patients with quantifiable urinary kappa or lambda chain concentration, a 50% reduction in daily light chain excretion (concentration x 24 hour urine volume). For patients with an elevated serum free light chain assay, reduction of 50% or more.
Time Frame: one year
Population: Participants who completed at least 3 cycles of treatment
Measure: Number; unit: participants
Arm/Group | Melphalan Revlimid and Dexamethasone
Number analyzed (Participants) | 14
participants | 7

2. Secondary Outcome: Number of Organs Improved or Stable Based on Description Below:
Description: Renal response - > 50% decrease in daily 24 hour proteinuria, without worsening renal insufficiency.
  Hepatic response - decrease of 2 centimeters or more of the liver span and/or decrease of the alkaline phosphatase by 50% if elevated at baseline.
  Cardiac response - decrease of 2 millimeters or more in mean left ventricular wall thickness in patients with baseline wall thickness > 11 mm or a decrease in New York Heart Association heart failure class.
  Autonomic nervous system response - resolution of orthostatic vital signs and symptoms, and resolution of symptoms of gastric atony or of functional ileus.
  Gastrointestinal response - a greater than one grade improvement in diarrhea due to biopsy proven amyloid.
  Peripheral nervous system response - resolution of clinical signs of peripheral neuropathy.
Time Frame: one year
Measure: Number; unit: number of organs stable or improved
Units Other Than Participants: involved organs
Arm/Group | Melphalan Revlimid and Dexamethasone
Number analyzed (Participants) | 14
Number analyzed (involved organs) | 24
number of organs stable or improved | 10

3. Secondary Outcome: Number of Participants Removed From Study Due to Toxicities
Description: Number of study participants removed from study treatment due to toxicities
Time Frame: One year
Population: All patients who have had at least one dose of drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Melphalan Revlimid and Dexamethasone
Number analyzed (Participants) | 16
Participants | 6

ADVERSE EVENTS:
Time Frame: 1 year
Description: Toxicity data was collected throughout study participation through 30 days after last dose.
Arm/Group | Melphalan Revlimid and Dexamethasone
Serious Adverse Events (participants affected / at risk) | 16/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan Revlimid and Dexamethasone (N=16)
thromboembolism (Blood and lymphatic system disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 2 (2)
heart failure (Cardiac disorders) | 4 (4)
infection (Infections and infestations) | 4 (4)
fatigue (General disorders) | 5 (5)
neutropenia (Blood and lymphatic system disorders) | 6 (6)
leukopenia (Blood and lymphatic system disorders) | 5 (5)
thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
anemia (Blood and lymphatic system disorders) | 2 (2)
pleural effusion - bilateral (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Elevated blood urea nitrogen test (Investigations) | 1 (1)
chest pressure (Cardiac disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
gout pain (Musculoskeletal and connective tissue disorders) | 1 (1)
pneumonia (Infections and infestations) | 2 (2)
sepsis (Infections and infestations) | 2 (2)
dehydration (Gastrointestinal disorders) | 1 (1)
septic shock (Infections and infestations) | 1 (1)
tear duct obstruction/infection (Eye disorders) | 1 (1)
increased creatinine (Investigations) | 2 (2)
gastrointestinal bleed (Gastrointestinal disorders) | 1 (1)
hypotension (Cardiac disorders) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
hyponatremia (Investigations) | 1 (1)
hyperglycemia (Investigations) | 1 (1)
pancytopenia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melphalan Revlimid and Dexamethasone (N=16)
abdominal bloating (Gastrointestinal disorders) | 2 (2)
abdominal cramping (Gastrointestinal disorders) | 2 (2)
altered taste (Gastrointestinal disorders) | 3 (3)
anemia (Blood and lymphatic system disorders) | 11 (24)
anorexia (Gastrointestinal disorders) | 4 (4)
anxiety (Psychiatric disorders) | 3 (3)
arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
aspiration (Gastrointestinal disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
blurring (Eye disorders) | 4 (4)
bradycardia (Cardiac disorders) | 1 (1)
chills (General disorders) | 3 (3)
cold intolerance (General disorders) | 2 (2)
confusion (Psychiatric disorders) | 2 (2)
congestive heart failure (Cardiac disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 9 (10)
cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
decreased bilirubin (Investigations) | 1 (1)
decreased iron (Investigations) | 1 (1)
decreased performance status (General disorders) | 2 (2)
decreased renal function (Renal and urinary disorders) | 1 (1)
depression (Psychiatric disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 5 (5)
dizziness (Nervous system disorders) | 6 (6)
dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
dry mouth (Gastrointestinal disorders) | 3 (3)
dysphagia (Gastrointestinal disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12)
dysuria (Renal and urinary disorders) | 1 (1)
early satiety (Gastrointestinal disorders) | 3 (3)
bruising (Skin and subcutaneous tissue disorders) | 5 (5)
edema (Blood and lymphatic system disorders) | 11 (13)
fatigue (General disorders) | 13 (14)
fever (General disorders) | 2 (2)
flatus (Gastrointestinal disorders) | 1 (1)
gout (Musculoskeletal and connective tissue disorders) | 3 (7)
headache (Nervous system disorders) | 3 (3)
hearing loss (Ear and labyrinth disorders) | 1 (1)
double vision (Eye disorders) | 1 (1)
hemorrhoida (Gastrointestinal disorders) | 2 (2)
hip fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 5 (5)
hyperglycemia (Investigations) | 7 (9)
hyperkalemia (Investigations) | 3 (5)
hypermagnesemia (Investigations) | 1 (1)
hypernatremia (Investigations) | 1 (1)
hyperphosphatemia (Investigations) | 1 (1)
hyperthyroidism (Endocrine disorders) | 2 (3)
hyperuricemia (Investigations) | 5 (5)
hypoalbuminemia (Investigations) | 6 (7)
hypocalcemia (Investigations) | 6 (6)
hypokalemia (Investigations) | 5 (5)
hypomagnesemia (Investigations) | 1 (1)
hyponatremia (Investigations) | 1 (1)
hypotension (Investigations) | 2 (3)
increased alkaline phosphatate (Investigations) | 3 (4)
increased Brain natriuretic peptide (Investigations) | 8 (8)
increased creatinine (Renal and urinary disorders) | 6 (7)
insomnia (General disorders) | 5 (5)
itchy eyes (Eye disorders) | 1 (1)
joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
leukocytosis (Blood and lymphatic system disorders) | 1 (1)
leukopenia (Blood and lymphatic system disorders) | 11 (13)
mental disturbance (Psychiatric disorders) | 1 (1)
mouth sores (Gastrointestinal disorders) | 1 (1)
hemorrhage (Gastrointestinal disorders) | 1 (1) — mucosal bleeding
muscle cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
peripheral neuropathy (Nervous system disorders) | 7 (9)
nocturia (General disorders) | 3 (3)
neutropenia (Blood and lymphatic system disorders) | 3 (4)
palpitations (Cardiac disorders) | 2 (2)
pancytopenia (Blood and lymphatic system disorders) | 2 (3)
polydipsia (Gastrointestinal disorders) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 2 (2)
hemorrhage (Gastrointestinal disorders) | 1 (1) — rectal bleed
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
sciatica (Nervous system disorders) | 1 (1)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
sweats (General disorders) | 3 (3)
thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
tinnitus (Ear and labyrinth disorders) | 4 (4)
infection (Infections and infestations) | 1 (1) — tooth abscess
tremors (Nervous system disorders) | 2 (2)
unsteady gait (Nervous system disorders) | 1 (1)
infection - upper respiratory (Infections and infestations) | 2 (5)
urinary frequency (Renal and urinary disorders) | 1 (1)
infection - urinary tract (Infections and infestations) | 2 (3)
vomiting (Gastrointestinal disorders) | 1 (1)
weakness (Nervous system disorders) | 6 (6)
weight loss (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes